CLINICAL TRIAL: NCT06989697
Title: Impact of Cilostazol and Ginkgo Leaf Extract on Cognitive Function in Elderly Patients With Type 2 Diabetes
Brief Title: Cilostazol-Ginkgo for Cognitive Function in Elderly Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Clinical Professor and Principal Investigator, Division of Endocrinology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B-2402-880-001
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabets Mellitus; Cognitive Ability, General
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol & Ginko Leaf Dried Ext. (Experimental): Renexin CR tab (cilostazol 200mg / Ginko Leaf Dried Ext. 160mg)
  Interventions: Drug: Cilostazol / Ginko Leaf Dried Ext.
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol / Ginko Leaf Dried Ext. — Patients will receive a light green, oval-shaped, sustained-release film-coated tablet containing a combination of cilostazol (200 mg) and ginkgo biloba extract (160 mg), administered orally once daily.
  Arms: Cilostazol & Ginko Leaf Dried Ext.
Drug: Placebo — Patients will receive a placebo identical in taste, aroma, and formulation to the active treatment, administered orally once daily.
  Arms: Placebo

SUMMARY:
This exploratory pilot study aims to evaluate the cognitive improvement effects of combination therapy with cilostazol (200 mg) and ginkgo biloba extract (160 mg) in elderly patients with type 2 diabetes mellitus. Both agents have demonstrated potential cognitive benefits through mechanisms such as enhanced cerebral blood flow, anti-inflammatory activity, and neuroprotection. Given the increased risk of cognitive decline and dementia in patients with type 2 diabetes, and the need for preventive strategies, this study will investigate whether the combination therapy can prevent or mitigate cognitive deterioration. Findings from this study may provide foundational data for the future development of therapeutic interventions targeting cognitive impairment in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes mellitus
* Adults aged 60 years or older
* Patients with a Mini-Mental State Examination (MMSE) score between 24 and 28 within the past 3 months

Exclusion Criteria:

* Patients with type 1 diabetes mellitus, diabetic ketoacidosis, or diabetic coma or precoma
* Patients with poorly controlled blood glucose (HbA1c > 10.0%)
* Patients with an MMSE score below 24
* Patients diagnosed with dementia (e.g., Alzheimer's disease)
* Patients with suspected cognitive impairment due to other causes
* Patients requiring antiplatelet or anticoagulant therapy other than the investigational product
* Patients with thyroid dysfunction requiring treatment (i.e., abnormal TSH levels)
* Patients with severe depression
* Patients with severe infections, recent surgery (perioperative status), or major trauma
* Patients with pituitary or adrenal insufficiency
* Patients with other medical conditions requiring hospitalization
* Patients with a history of alcohol or drug abuse within 1 year prior to screening
* Patients with a history of taking medications that may affect cognitive function within 3 months prior to screening
* Patients deemed by the investigator to be otherwise unsuitable for study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) Score From Baseline to 6 Months | 6 months
  The MMSE is a widely used test of cognitive function among the elderly. It includes tests of orientation, attention, memory, language, and visual-spatial skills. Scores range from 0 to 30, with higher scores indicating better cognitive function. A change in total MMSE score from baseline to 6 months will be assessed.

SECONDARY OUTCOMES:
Change in Korean Dementia Screening Questionnaire (KDSQ) Score From Baseline to 6 Months | 6 months
  The Korean Dementia Screening Questionnaire (KDSQ) is a caregiver- or self-administered tool used to screen for cognitive decline in older adults. It consists of 15 items, each scored from 0 to 2, for a total possible score of 0 to 30.
  Higher scores indicate greater cognitive impairment. A change in the total KDSQ score from baseline to 6 months will be assessed.
Change in Korean Version of the Montreal Cognitive Assessment (K-MoCA) Score From Baseline to 6 Months | 6 months
  The K-MoCA is a cognitive screening tool used to detect mild cognitive impairment and early dementia (https://mocacognition.com/paper/). It assesses multiple domains including attention, executive function, memory, language, visuospatial skills, abstraction, calculation, and orientation.
  Higher scores indicate better cognitive function (Score Range: 0 to 30). A change in the total K-MoCA score from baseline to 6 months will be assessed.
Change in Global Deterioration Scale (GDS) Stage From Baseline to 6 Months | 6 months
  The GDS is a clinical tool used to assess the severity of cognitive decline, particularly in Alzheimer's disease and other dementias. It includes 7 stages, ranging from:
  Stage 1: No cognitive decline ~ Stage 7: Very severe cognitive decline. Higher scores indicate more severe cognitive impairment. A change in the GDS stage from baseline to 6 months will be recorded based on clinical assessment.
Change in Short Form-36 Health Survey (SF-36) Scores From Baseline to 6 Months | 3, 6 months
  The SF-36 Health Survey is a 36-item, patient-reported questionnaire that assesses health-related quality of life across 8 domains:
  Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Problems, Energy/Fatigue (Vitality), Emotional Wellbeing (Mental Health), Social Functioning, Pain (Bodily Pain), General Health Perceptions.
  Each domain is scored separately on a scale from 0 to 100, with higher scores indicating better health status. Summary scores, such as the Physical Component Summary (PCS) and Mental Component Summary (MCS), may also be calculated.
  Changes in domain and/or summary scores from baseline to 6 months will be assessed.

OTHER OUTCOMES:
Glucose regulation | 3, 6 months
  Change in HbA1c level From Baseline to 6 Months
Lipid Panel | 3, 6 months
  Change in Lipid Profile From Baseline to 6 Months
Renal Function | 3, 6 months
  Change in estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) from baseline to 6 Months
Liver Function | 3, 6 months
  Change in Liver Function (AST, ALT) From Baseline to 6 Months
C-Reactive Protein | 6 months
  Change in hsCRP Levels From Baseline to 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided